CLINICAL TRIAL: NCT05995795
Title: Arthroscopic Release Of Shoulder Internal Rotation Contracture In Brachial Plexus Palsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hamed Mohamed, DR.mohamed hamed, Assiut University
Other Study IDs: Arthroscopy in OBBP
Record Dates: First submitted 2023-05-10; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Arthroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ARTHROSCOY — arthroscopy

SUMMARY:
The purpose of this study is to evaluate the efficacy periarticular capsuloligamentous arthroscopic release of shoulder internal rotation contracture in brachial plexus palsy without any further intervention as tendon transfer.

DETAILED DESCRIPTION:
Obstetrical brachial plexus paralysis (OBPP) refers to complete or partial injury of the brachial plexus produced at the time of birth. OBPP involves most commonly the upper cervical roots (C5, C6) resulting in muscle imbalance between internal and external rotators of the shoulder . Although the majority of the patients (80-90%) recover spontaneously, some have a remaining imbalance causing severe functional impairment . In addition to diminished function, prolonged muscle contractures result in bony deformities in both the glenoid and proximal humerus. Internal rotation contractures due to external rotational weakness are the most common deformity in OBPP. Contracture release, tendon transfers, and rotational osteotomies are surgical methods used, depending on the level of deformity and the patient's age. To achieve functional external rotation of the arm, contracted structures should be released first. Currently, there is a lack of consensus on which procedures over the best outcome for mobility and function, and what are the precise indications for each type of surgery. There is also a large variation of practice between centers

ELIGIBILITY:
Inclusion Criteria:

* children from 1 year to 15years of age.
* all genders
* patients with brachial plexus injury operated or not with internal rotation contracture
* patient with traumatic brachial plexus injury have residual internal rotation contracture

Exclusion Criteria:

* History of septic shoulder
* Flail anaethetic limb
* glenohumeral posterior sublaxation or dislocation in CT

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with brachial plexus injury operated or not with internal rotation contracture
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with failure of initial intervention | 1 year
  change of improvement of passive and active external rotation of operated shoulder using mallet score

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Koteb, phD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hale HB, Bae DS, Waters PM. Current concepts in the management of brachial plexus birth palsy. J Hand Surg Am. 2010 Feb;35(2):322-31. doi: 10.1016/j.jhsa.2009.11.026. PMID 20141905